CLINICAL TRIAL: NCT05401253
Title: The Association of Different Levels of Physical Activity on Postoperative Pulmonary Complications in Patients Undergoing Thoracoscopic Lung Resection Surgery: A Prospective Cohort Study
Brief Title: The Association of Different Levels of Physical Activity on Postoperative Pulmonary Complications in Patients Undergoing Thoracoscopic Lung Resection Surgery
Status: Completed | Type: Observational
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Changping Gu, Professor, Qianfoshan Hospital
Other Study IDs: YXLL-KY-2022(014)
Record Dates: First submitted 2022-04-25; First posted 2022-06-02 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pulmonary Complications
Keywords: Postoperative pulmonary complications; Lung resection surgery; Physical activity; General anesthesia
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial blood samples from patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adequate physical activity group: At least 600 met-minutes /week for five or more days of walking, moderate and strenuous physical activity per week.
- Insufficient physical activity group: Less than 600 met-minutes /week for five or more days of walking, moderate and strenuous physical activity per week.

SUMMARY:
This study aimed to predict different physical activity (PA) levels in patients undergoing thoracoscopic lung resection surgery (LRS) using the International Physical Activity Questionnaire (IPAQ) and investigate the association between the PA levels and the incidence of postoperative pulmonary complications (PPCs). The patients were classified into the high-level and low-level PA groups based on the IPAQ scores. The incidence of PPCs within postoperative 5 days, number of PPCs, the incidence of postoperative adverse events (PAEs) within postoperative 5 days, extubation time, length of hospital stay (LOS), unplanned admission to the intensive care unit (ICU), and the mortality 1-month postoperatively were recorded. Arterial blood samples were collected before induction of anesthesia and 1 hour postoperatively, and the supernatants were centrifuged for cytokine analysis. Binomial logistic analysis was performed to determine the relationship between predefined variables and PPCs. Receiver operating characteristic (ROC) curve analysis was performed to identify independent risk factors, and the area under the curve (AUC) was calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years and younger than 80 years;
2. Patients scheduled to accept elective thoracic surgery under general anesthesia;
3. Patients of American Society of Anesthesiologists (ASA) Ⅱ～Ⅲ level grade;
4. Patients signed the informed consent form for the clinical study.

Exclusion Criteria:

1. Patients with moderate or severe chronic obstructive pulmonary disease (GOLD Grade III or IV level grade)；
2. Patients with severe or uncontrolled bronchial asthma；
3. Patients with severe neuromuscular disease or thoracic malformation；
4. Patients with severe heart disease (New York Heart Association Class III or IV level grade or acute coronary syndrome or persistent ventricular arrhythmia)；
5. Patients with cognitive dysfunction；
6. Patients who have participated in other clinical trials within the previous 30 days；
7. Patients with coagulation dysfunction；
8. Patients who received radiotherapy or chemotherapy within 2 months before surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18~80 years undergoing elective thoracoscopic lung resection surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Incidence of pulmonary complications | Within five days after surgery
  1. Respiratory Infection
  2. Respiratory Failure
  3. Pleural Effusion
  4. Atelectasis
  5. Pneumothorax
  6. Bronchospasm
  7. Aspiration pneumonitis

SECONDARY OUTCOMES:
The arterial levels of inflammatory markers | before induction of anesthesia(T0),1.5 hours after the beginning of surgery(T2),3 hours after the beginning of surgery(T3)and 1 hour after the end of surgery(T4).
  interleukin-6(IL-6), interleukin-8(IL-8), tumor necrosis factor-α(TNF-α)
The number of postoperative pulmonary complications | Within five days after the surgery
Extubation time | The time from the end of surgery to the removal of the endotracheal intubation.
Postoperative length of stay | During the study procedure
Incidence of postoperative adverse events | Within five days after operation
  1. arrhythmia
  2. acute cardiovascular disease (myocardial infarction, heart failure)
  3. acute cerebrovascular disease (cerebral infarction, cerebral hemorrhage, TIA)
  4. acute postoperative psychiatric disorder (delirium,somnolence,coma)
  5. shock
Unplanned admission to the ICU | Within five days after operation
Mortality 1 month after surgery | Within 1 month of the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Changping Gu, doctor, Principal Investigator — Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University
Locations (1):
- China, Shandong Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qiu L, Zhao L, Wang B, Yang L, Cao C, Lv M, Xu M, Hou M, Wang X, Wang Y, Gu CP. Predicting the association of different levels of physical activity on postoperative pulmonary complications using the international physical activity questionnaire in patients undergoing thoracoscopic lung surgery under general anaesthesia: protocol for a prospective cohort study. BMJ Open. 2024 May 15;14(5):e077183. doi: 10.1136/bmjopen-2023-077183. PMID 38749692